CLINICAL TRIAL: NCT03286465
Title: Pilot, Randomized Trial of the Use of Pediatric Size Phlebotomy Tubes in Adult Critically Ill Patients to Reduce Red Blood Cell Transfusions
Brief Title: Use of Pediatric Size Phlebotomy Tubes in Adult Critically Ill Patients to Reduce Red Blood Cell Transfusions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Javier Barreda Garcia, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSC-MS-17-0280
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Results first posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Anemia
Keywords: blood transfusion
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Pediatric phlebotomy tubes (Experimental): Use of pediatric size tubes for diagnostic blood collection.
  Interventions: Device: Pediatric phlebotomy tubes
- Adult phlebotomy tubes (Active Comparator): Use of adult size tubes for diagnostic blood collection.
  Interventions: Device: Adult phlebotomy tubes

INTERVENTIONS:
Device: Pediatric phlebotomy tubes — Use of pediatric size tubes for diagnostic blood collection.
  Arms: Pediatric phlebotomy tubes
Device: Adult phlebotomy tubes — Use of adult size tubes for diagnostic blood collection.
  Arms: Adult phlebotomy tubes

SUMMARY:
This study will evaluate the hypothesis that the use of pediatric size phlebotomy tubes reduces red blood cell (RBC) transfusions in adult intensive care unit (ICU) patients compared with the use of adult size tubes.

ELIGIBILITY:
Inclusion Criteria:

* New admission to the medical or transplant ICU at Memorial Hermann Hospital in Houston
* ICU admission hemoglobin level of at least 7 g/dL. The ICU admission hemoglobin will be the most recent hemoglobin value available at the time of screening for inclusion in the study.
* Randomization is expected within 12 hour of admission to the ICU

Exclusion Criteria:

* Clinical bleeding. Defined as menstrual bleeding, bleeding leading to a change in the frequency of hemoglobin monitoring or to an order for a medication, transfusion, procedure, or consultation intended to prevent or treat bleeding.
* Known hemolytic disorder (e.g. sickle cell disease, hereditary spherocytosis, autoimmune hemolytic anemia)
* Bone marrow disorder (e.g. aplastic anemia, marrow infiltration disorder, chemotherapy within the last 8 weeks)
* Jehovah's Witnesses
* Patient is comfort care measures only
* Refractory shock: mean arterial blood pressure below 60 mmHg despite maximal doses of 3 vasopressors. Maximal dose of vasopressors are as follows: Norepinephrine 70 mcg/min; vasopressin 0.04 units/min; epinephrine 35 mcg/min; dopamine 20 mcg/kg/min; phenylephrine 350 mcg/min
* Severe acidosis: potential of hydrogen (pH) below 7 in more than one arterial blood gas within 24 hours of ICU admission in the absence of diabetic ketoacidosis Surgical admission diagnosis
* Pregnancy
* Current prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Barreda Garcia, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States

REFERENCES:
- [Derived] Barreda Garcia J, Xian JZ, Pedroza C, Salahuddin M, Mak G, Keene A, Cherian SV, Young AY, Vijhani P, Doshi PB. Pediatric size phlebotomy tubes and transfusions in adult critically ill patients: a pilot randomized controlled trial. Pilot Feasibility Stud. 2020 Aug 8;6:112. doi: 10.1186/s40814-020-00657-3. eCollection 2020. PMID 32782818

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pediatric Phlebotomy Tubes | Adult Phlebotomy Tubes
Started | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pediatric Phlebotomy Tubes | Adult Phlebotomy Tubes | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (16.7) | 57 (18.5) | 56.2 (17.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 51 | 96
  Male | 55 | 49 | 104
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 36 | 46 | 82
  White | 38 | 39 | 77
  Other | 26 | 15 | 41
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 100 | 100 | 200
Hemoglobin concentration at intensive care unit (ICU) admission [Mean (Standard Deviation); unit: g/dL] | 11.4 (2.4) | 11.1 (2.3) | 11.24 (2.35)
Time from ICU admission to randomization [Median (Inter-Quartile Range); unit: hours] | 5.3 [1.5 to 8] | 5.7 [2.6 to 8.6] | 5.64 [2.15 to 8.47]
Estimated blood volume [Median (Inter-Quartile Range); unit: liters] | 4.9 [4.2 to 5.6] | 4.6 [3.9 to 5.4] | 4.77 [3.97 to 5.51]
Number of participants with chronic hemodialysis [Count of Participants; unit: Participants] | 12 | 12 | 24
Number of participants with chronic kidney disease but no dialysis [Count of Participants; unit: Participants] | 13 | 11 | 24
Number of participants with active malignancy [Count of Participants; unit: Participants] | 5 | 5 | 10
Number of participants with recent history of anemia [Count of Participants; unit: Participants] | 45 | 47 | 92
Charlson comorbidity index [Median (Inter-Quartile Range); unit: score on a scale] — The Charlson comorbidity index predicts 10-year survival in patients with multiple comorbidities. Total score rantes from 0 to 33. The higher the score, the higher the chance of mortality.
  score on a scale | 3.0 [2 to 6] | 4.0 [2 to 5] | 3 [2 to 6]
ICU Admission Diagnosis [Count of Participants; unit: Participants]
  Infection | 55 | 46 | 101
  Acute Cardiovascular Disorder | 21 | 24 | 45
  Acute renal failure | 40 | 31 | 71
  Metabolic disorder | 32 | 36 | 68
  Non-infectious inflammatory disorder | 19 | 11 | 30
  Other | 22 | 31 | 53
Number of participants who had invasive mechanical ventilation [Count of Participants; unit: Participants] | 50 | 51 | 101
APACHE II score [Median (Inter-Quartile Range); unit: score on a scale] — The APACHE II score estimates ICU mortality. Total score ranges from 0 to 71 points, with higher scores indicating greater mortality.
  score on a scale | 22.0 [14 to 29] | 23.0 [16 to 28] | 22 [15.75 to 28.25]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Hemoglobin Less Than 7 g/dL or Red Blood Cell (RBC) Transfusion Order
Time Frame: from time of admission to intensive care unit (ICU) to 30 days after admission to ICU
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Phlebotomy Tubes | Adult Phlebotomy Tubes
Number analyzed (Participants) | 100 | 100
Participants | 6 | 11

2. Secondary Outcome: Rate of Change in Hemoglobin (g/dL/Day) While in the Intensive Care Unit (ICU)
Description: This will be calculated as the most recent hemoglobin prior to randomization minus the last hemoglobin prior to ICU discharge, death, RBC transfusion, clinical bleeding, surgery, or change of clinical status to comfort measures, divided by the number of days (rounded to the nearest 0.5) between these two values (crude estimate).
Time Frame: from time of randomization to completion of study (up to 30 days after ICU admission)
Measure: Median (Inter-Quartile Range); unit: g/dL/day
Arm/Group | Pediatric Phlebotomy Tubes | Adult Phlebotomy Tubes
Number analyzed (Participants) | 100 | 100
g/dL/day | -0.21 [-0.48 to 0.021] | -0.2 [-0.54 to 0.038]

3. Secondary Outcome: Number of Participants Who Received a Red Blood Cell (RBC) Transfusion While in the ICU
Time Frame: completion of study (up to 30 days after ICU admission)
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Phlebotomy Tubes | Adult Phlebotomy Tubes
Number analyzed (Participants) | 100 | 100
Participants | 4 | 9

4. Secondary Outcome: Number of Participants With at Least One Inadequate Blood Sample for Laboratory Analysis
Description: An inadequate blood sample is defined as any blood sample that requires recollection.
Time Frame: completion of study (up to 30 days after ICU admission)
Population: This outcome data was not collected in the arm using adult phlebotomy tubes.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Phlebotomy Tubes | Adult Phlebotomy Tubes
Number analyzed (Participants) | 100 | 0
Participants | 7 |

5. Secondary Outcome: ICU Mortality
Time Frame: completion of study (up to 30 days after ICU admission)
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Phlebotomy Tubes | Adult Phlebotomy Tubes
Number analyzed (Participants) | 100 | 100
Participants | 9 | 10

6. Secondary Outcome: Total Phlebotomy Volume
Description: The total phlebotomy volume is the total volume of blood collected over all days and is estimated based on the maximum volume needed for each type of blood test, as follows. In the pediatric tube arm, the volumes were 0.5 milliliters (mL) for hematology, 0.6 mL for chemistries (plasma), and 2.5 mL for coagulation tests. In the adult tube group, the volumes were 5.5 mL for hematology, 5 mL for chemistries (plasma), and 3.8 mL for coagulation. In both arms, tube volumes for lactate, immunology (serum), arterial blood gases, and blood cultures were 5 mL, 6.5 mL, 1 mL, and 10 mL, respectively.
Time Frame: completion of study (up to 30 days after ICU admission)
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Pediatric Phlebotomy Tubes | Adult Phlebotomy Tubes
Number analyzed (Participants) | 100 | 100
mL | 21 [7 to 38] | 50 [27 to 100]

ADVERSE EVENTS:
Time Frame: time of randomization to completion of study (up to 30 days after ICU admission)
Description: Systematically assessed for RBC transfusion-related adverse events.
Arm/Group | Pediatric Phlebotomy Tubes | Adult Phlebotomy Tubes
All-Cause Mortality (participants affected / at risk) | 9/100 | 10/100
Serious Adverse Events (participants affected / at risk) | 9/100 | 10/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pediatric Phlebotomy Tubes (N=100) | Adult Phlebotomy Tubes (N=100)
death (General disorders) | 9 (9) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-28): https://cdn.clinicaltrials.gov/large-docs/65/NCT03286465/Prot_SAP_000.pdf